CLINICAL TRIAL: NCT01573650
Title: Optimization of Peripheral Nerve Reconstruction: A Non-inferiority Trial
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Version 2, 01/04/2012
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Peripheral Nerve Injury Digital Nerve Hand Left

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group 1: Group 1a (standard): Epineural Suture Group 1b (experimental): Epineural suture and Fibrin Wrap
- group 2: Group 2a (standard): Epineural suture and autologous nerve transplantation from lateral antebrachial cutaneous nerve (LACN) Group 2b (experimental): Epineural suture and Fibrin Conduit

SUMMARY:
1. To analyse the outcome of different treatment options of peripheral nerve repair with no gap (group 1) and with a critical sized (>5mm) defect (group 2) in order to optimize peripheral nerve repair
2. To reduce morbidity with the same outcome

DETAILED DESCRIPTION:
Patients planned to undergo peripheral nerve repair after traumatic nerve injury with either no gap (group 1) or with a critical sized defect (>5mm, group 2) of the finger providing written informed consent to this investigation will be randomised in two groups:.

Group 1: nerve repair with no gap Group 1a (standard): Epineural Suture Group 1b (experimental): Epineural Suture and Fibrin Wrap Group 2: Nerve repair with a critical sized (>5mm) defect Group 2a (standard): Epineural suture and autologous nerve transplantation from lateral antebrachial cutaneous nerve (LACN) Group 2b (experimental): Epineural suture and Fibrin Conduit

In all groups an epineural suture will be performed (suture enhancement). The outcome of fibrin enwrapment and fibrin conduit will be compared to the standard treatment option to date (direct nerve repair and autologous nerve graft, respectively). Randomization will be performed using a computer-base algorithm (www.randomizer.at). Ambulatory follow up of patients is carried out by the Department of Plastic, Reconstructive and Aesthetic Surgery, Handsurgery, University Hospital Basel. The outcome-assessor as well as the patient will be blinded for analysis and the outcome-assessor will have no access to the surgery report.

The investigator's aim is to analyse 48 patients within 12 months. Since 100 patients undergo peripheral nerve repair annually in the Department of Plastic, Reconstructive and Aesthetic Surgery, Handsurgery at the University Hospital Basel, patient accrual appears unproblematic.

After completion, statistical analysis focusing on the comparison of the different types of surgery concerning the clinical parameters 2-Point Discrimination (PD), Semmes Weinstein test, and electroneurography will be conducted.

After six months, no difference will be expected between group 1a and 1b or 2a and 2b, respectively. In the investigator's experience there will be no confounders which may influence nerve regeneration. A similar patient satisfaction will be expected between the groups. The investigator expect a higher patient satisfaction in group 2b than in group 2a due to nerve tissue harvest. Between group 1a and 1b no difference is expected regarding MHQ.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic peripheral nerve injury of the finger(s) who are to be treated with peripheral nerve repair at the Department of Plastic, Reconstructive and Aesthetic Surgery, Handsurgery, University Hospital of Basel
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Age > 90 years
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic peripheral nerve injury of the finger(s) who are to be treated with peripheral nerve repair at the Department of Plastic, Reconstructive and Aesthetic Surgery, Handsurgery, University Hospital of Basel Written informed consent
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
2-PD | 2wks, 3mts and 6mts

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kalbermatten, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland